CLINICAL TRIAL: NCT00118391
Title: Enhanced Cognitive Behavior Therapy for the Treatment of Pathological Gambling
Brief Title: Cognitive-Behavioral Treatment of Gambling
Acronym: CBT/CM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Nancy Petry, PhD, University of Connecticut Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH060417-02 (NIH); R01MH060417-02 (NIH)
Record Dates: First submitted 2005-07-06; First posted 2005-07-11 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Gambling; Mental Health
Keywords: Pathological Gambling; CBT; CM
MeSH Terms: conditions — Gambling; Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — Receive 8 50-minute sessions of one-on-one cognitive behavioral therapy
Behavioral: Contingency management — Receive vouchers that can be spent on rewards for completing activities that support abstinence from gambling

SUMMARY:
This study will determine the effectiveness of cognitive behavior therapy (CBT) and contingency management (CM) in reducing gambling behaviors and other related problems in pathological gambling.

Study hypothesis: Participants who receive CBT and CM will attend more treatment sessions and show better outcomes than those who receive CBT alone.

DETAILED DESCRIPTION:
Pathological gambling has become an increasingly problematic condition in the United States, often causing serious financial, psychological, and public health consequences. In an effort to treat this growing problem, researchers have evaluated numerous therapies; one such therapy is CBT. CBT has been shown to improve pathological gambling outcomes. However, evidence suggests that adding CM to CBT could result in even more improved outcomes. This study will compare the effectiveness of CBT and CM with that of CBT alone in reducing pathological gambling.

This study will last 12 months. Participants will be randomly assigned to receive either CBT and CM or CBT alone for 8 weeks. CBT will focus on reducing gambling urges and helping patients develop alternative behaviors to gambling. CM will focus on encouraging patients to avoid gambling. Participants in the CBT and CM group will receive voucher incentives for completing homework assignments and engaging in non-gambling social activities. The vouchers will allow participants to take part in non-gambling activities of their choice. Changes in gambling activities and problems will be assessed with self-report scales and interviews at study start and at Weeks 10, 24, and 52.

Participants will be asked to identify at least one person who knows about their gambling and will have regular contact with them over the 12 months of the study. This person will be interviewed at study start and at Months 2, 6, and 12. Contact persons will be asked about participants' gambling behaviors, personal relationships, legal problems, use of health care and mental health services, and how the participant can be contacted if he or she moves.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00158314

http://clinicaltrials.gov/show/NCT00618462

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pathological gambling
* At least 1 gambling episode within 30 days prior to study entry
* Able to read English at a 5th grade level
* Willing and able to comply with all study requirements

Exclusion Criteria:

* Uncontrolled psychiatric conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-11; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Addiction Severity Index (ASI) gambling severity scores
amount spent gambling per gambling episode
longest period of non-gambling
days until first gambling episode
percent of days gambling
proportion meeting diagnostic criteria
number of treatment sessions attended

SECONDARY OUTCOMES:
Psychosocial functioning

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M. Petry, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States